CLINICAL TRIAL: NCT02480283
Title: Chronic Cannabis Smoking, Oxidative Stress and the Pulmonary Innate Immune Response
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 14-1957; UL1TR001082 (NIH)
Record Dates: First submitted 2015-05-27; First posted 2015-06-24 (Estimated); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Cannabis Smoking; Oxidative Stress
MeSH Terms: conditions — Marijuana Smoking | interventions — Bronchoscopy; X-Rays; Phlebotomy; Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 1. Urine
  2. Exhaled Breath Condensate
  3. Blood/Plasma
  4. Bronchial brushings
  5. Bronchoalveolar Lavage
  6. Oral rinse
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control: Subjects aged 18 to 55 who have never used cannabis by self report (validated via urine drug screen), who have never used tobacco/cigarettes and have the capacity to give informed consent.
  Interventions: Procedure: Bronchoscopy; Radiation: Chest X-ray; Procedure: Venipuncture; Procedure: Intravenous Catheter
- Cannabis Smokers: The exposed cohort will have daily or near daily cannabis smoking histories equivalent to a minimum of 20 joint years (number of joints smoked per day multiplied by years of cannabis smoking), will not have a significant tobacco/cigarette smoking history and will be able to provide informed consent.
  Interventions: Procedure: Bronchoscopy; Radiation: Chest X-ray; Procedure: Venipuncture; Procedure: Intravenous Catheter

INTERVENTIONS:
Procedure: Bronchoscopy — Passage of a thin flexible tube through the mouth, into the windpipe and then into the bronchial tubes so that the study doctor can look into the lungs to perform Bronchoalveolar lavage (BAL), cytologic brushing, and protected specimen brushing.
Radiation: Chest X-ray — To identify any previously undiagnosed lung disease that will either increase the risk of bronchoscopy or confound results of the study.
  Other Names: CXR
Procedure: Venipuncture — To collect blood cells and serum for analyses.
  Other Names: Blood Test
Procedure: Intravenous Catheter — To administer the appropriate medications for the bronchoscopy procedure.
  Other Names: IV

SUMMARY:
This study plans to evaluate the effects of chronic cannabis smoking on lung health by evaluating its effects on pulmonary health, lung physiology and alveolar macrophage function.

DETAILED DESCRIPTION:
I. Hypotheses and Specific Aims:

With changing legislation, the landscape of cannabis use is shifting; data demonstrates that public perception of marijuana's "safety" has contributed to increasing usage most commonly via the inhaled route (smoking). The effects of habitual cannabis smoking on lung health, however, remains unclear. Spirometric data has been inconclusive regarding risk of airflow limitation and development of chronic obstructive pulmonary disease, a finding that may be attributable to inaccurate reporting due to its former illegal nature. It seems clear, however, that these patients suffer from an increased incidence of bronchitis symptoms from an uncertain pathophysiologic mechanism. Animal data from the 1990s demonstrates that cannabinoid exposure (of which Tetrahydrocannabinol (THC) is an example) results in increased intra-pulmonary oxidative stress indices and immunomodulatory effects resulting in abnormal macrophage function; a finding that may be related the aforementioned symptoms. However, this data is likely now outmoded given the markedly increased (THC) content of today's cannabis for sale (12 percent Tetrahydrocannabinol (THC) compared to 3 percent in the 1990s). Furthermore, most of these findings have not been validated in human subjects. Thus, the investigators hypothesize that habitually smoked cannabis increases intrapulmonary oxidative stress resulting in impaired alveolar macrophage (AM) phagocytosis, elicits an attenuated AM response to pathogen-associated molecular patterns (PAMPs) and promotes AM apoptosis thereby increasing risk of upper and lower airway infections.

II. Background and Significance:

Cannabis use in the United States is rising since legalization for medical and, more recently, recreational purposes. The United Nations Office on Drugs and Crime estimates that in 2012, when cannabis was legal for medical purposes in 17 states, but illegal for recreational consumption nationally, cannabis use among the American population increased from 11.5% to 12.1%. Over the past 2 years, an additional seven states have legalized medical cannabis, and Colorado and Washington have recently legalized its sale for recreational use. Since January 2014, publicly available Colorado data indicate increasing tax revenue from cannabis sales (both medical and recreational), suggesting a rise in state-wide consumption in a relatively short period of time.

Effects of modern inhaled cannabis on lung health are not established. Published epidemiologic data collected prior to the widespread legalization of cannabis and commercialization of the cannabis industry demonstrate consistent associations between "regular" (e.g. near daily) and "heavy" (e.g. for multiple years) cannabis use with poorer lung health. Clinically, regular inhaled cannabis users complain of increased chronic bronchitis symptoms (eg. wheeze, chronic cough) compared to non-smokers; an increased use of medical services for respiratory infections due to immunosuppressive effects of the drug has also been reported. However, characterization of cannabis use in these investigations varies widely, ranging from 7 joint-years (1 joint per day for 1 year) 12 to 117 joint-years in cohorts examined. These studies were also potentially confounded by under-reporting of cannabis use due to the drug's illegal status, and concomitant use of inhaled tobacco in some study populations. Moreover, the quantity of THC in modern cannabis products has been increasing over the past two decades. Therefore, it remains unclear what use patterns of modern inhaled cannabis are harmful to lung health, although more cannabis is being consumed now than ever before, both for medical and recreational purposes. Today, due to the decriminalization of cannabis sale and purchase, the accuracy of self-reported cannabis use is likely much greater than in prior investigations, providing a novel opportunity to more accurately establish patterns of use associated with ill effects on health. Importantly, no study to date has utilized time series analyses, such as the time line follow-back (TLFB), to quantitate the effects of regular cannabis consumption in association with lung health. TLFB techniques are used extensively to quantitate substance use among chronic users of alcohol, tobacco, and more recently, cannabis. TLFB are calendar-assisted, structured interviews that cue memory to enhance accurate recall, and have been determined to be both reliable and valid in quantitating current substance use in detail. TLFB interviews to characterize past 30 day cannabis use have been routinely conducted in research subjects by Dr. Corsi's (co-mentor to Dr. Biehl) research group since 2010, and longer term joint-year data has been collected as well.

Inhaled cannabis use adversely affects function of alveolar macrophages (AMs), critical pulmonary innate immune effectors. AMs express cannabinoid (CB) receptors, primarily CB2, on their surface, whose ligand is THC15 (a cannabinoid). AMs represent the first line of defense against invading pathogens in the lower airways, and function to keep the lungs sterile. Published investigations using AMs isolated via bronchoalveolar lavage (BAL) from small numbers (n<20) of habitual inhaled cannabis users have reported an inappropriately diminished response to S. aureus, an important lung pathogen. When AMs were exposed to S. aureus, they exhibited decreased bacterial phagocytosis and killing; hampered production of the pro-inflammatory cytokines tumor necrosis factor-α, IL-6, and granulocyte monocyte colony stimulating factor; and decreased production of nitric oxide. Preclinical data has suggested that AM viability and apoptosis may also be adversely influenced by THC in a dose- and time-dependent manner through the CB2 receptor, further impairing the AM's ability to respond to pathogens. As mentioned, cannabis use is increasing on a per capita basis, and continues to be used via an inhaled route, while its THC quantity is increasing. Collectively, this suggests the possibility that individuals who regularly use small doses of inhaled cannabis, or have used cannabis for a shorter length of time, may still be at risk for AM dysfunction, clinically manifested by increased respiratory symptoms and an increased risk for pulmonary infections, particularly since pre-clinical data has consistently reported adverse effects of cannabis exposure on infectious disease resistance.

Cannabis exposure in vitro leads to oxidative stress that in turn affects pulmonary cellular viability. Murine lung epithelial cells exposed to cannabis smoke extract in vitro demonstrate a dose-related increase in oxidative stress, while human lung BEAS-2B cells exposed to cannabis smoke extract in vitro display an increase in reactive oxygen species production. Enhanced oxidative stress in each investigation was further associated with evidence of cytotoxicity, characterized by cellular apoptosis and DNA damage. It seems possible, then, that enhanced oxidative stress due to habitual inhaled cannabis may additionally influence the viability and function of AMs in the lower airways. However, the effect of inhaled cannabis on oxidative stress and its relationship to AMs has never been specifically explored with primary cells from human subjects.

In summary, our collaboration will utilize validated methods to characterize regular and chronic cannabis use patterns among exclusive medical and/or recreational cannabis users, in order to examine their impact on cells critical to the maintenance of lung health. Information the investigators derive may be used to counsel active and contemplating cannabis users, and inform medical providers and researchers.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA for CANNABIS USING patient: Subjects will be eligible if they meet ALL of the following criteria:

1. Daily or near daily cannabis use (inhaled via joint/cigarette or pipe) equivalent to AT LEAST 20 "joint years" (number of joints/cigarettes per day multiplied by number of years during which cannabis was smoked) by self-report and validated through urine drug screen.
2. Never or limited exposure to inhaled tobacco products (equivalent to LESS THAN one "pack year" in a lifetime) by selfreport and validated through negative urine cotinine screen.
3. Capacity to answer screening questions and provide informed consent at time of interview, along with contact information

INCLUSION CRITERIA for CONTROL patient: Subjects will be eligible if they meet all of the following:

1. No cannabis use ever by self-report, and validated through urine drug screen.
2. Never users of tobacco/cigarettes
3. Capacity to answer screening questions and provide informed consent at time of interview, along with contact information.

Exclusion Criteria:

EXCLUSION CRITERIA for CANNABIS USING patient: Subjects will be ineligible if they meet ANY of the following criteria:

1. LESS THAN near daily cannabis use (inhaled via joint/cigarette or pipe) equivalent to LESS THAN 20 "joint years" (number of joints/cigarettes per day multiplied by number of years during which cannabis was smoked) or a negative urine drug screen (for cannabis)
2. Inhaled tobacco product exposure EXCEEDING one "pack year" or a positive urine cotinine screen
3. Elevated AUDIT-C score: A 3 item questionnaire to identify subjects with alcohol use disorders.
4. Prior medical history of liver disease: cirrhosis, total bilirubin > 2.0 mg/dL or albumin <3
5. Prior medical history of myocardial infarction or congestive heart failure
6. Prior medical history of end-stage renal disease or serum creatinine >3 mg/dL
7. Prior history of or current use of illicit drug use defined as a positive toxicology screen for opiates or cocaine
8. Prior history of diabetes mellitus
9. Prior history of chronic obstructive pulmonary disease (COPD) or asthma that is not clinically controlled (have not required systemic corticosteroids in the past month)
10. Prior history of HIV, not controlled or on medication
11. Peripheral white blood cell count of less than 3000
12. Acute worsening (<7 days) in respiratory symptoms (such as change in cough frequency or sputum production, fever, dyspnea, abnormal chest radiograph), or room air pulse oximetry of < 92% at rest or spirometry of < 50% predicted for FEV1 and FVC
13. Use of systemic antibiotics for any reason in the past month (4 weeks)
14. Failure of a subject or the subject's substance abuse counselor to provide assent
15. Nutritional risk index of less than 95
16. Age < 21 or > 55 (using an age of 55 limits the likelihood of comorbid conditions that may increase the risk of adverse events with bronchoscopy)
17. Pregnancy
18. Decisionally challenged
19. Prisoners.

EXCLUSION CRITERIA for CONTROL patient: Subjects will be ineligible to participate if they meet ANY of the following criteria:

1. History of inhaled cannabis exposure EXCEEDING one "joint year" or positive urine toxicology screen (for cannabis)
2. History of inhaled tobacco product exposure EXCEEDING one "pack year" or a positive urine cotinine screen
3. Elevated AUDIT-C score: A 3 item questionnaire to identify subjects with alcohol use disorders.
4. Prior medical history of liver disease: cirrhosis, total bilirubin > 2.0 mg/dL or albumin <3
5. Prior medical history of myocardial infarction or congestive heart failure
6. Prior medical history of end-stage renal disease or serum creatinine >3 mg/dL
7. Prior history of or current use of illicit drug use defined as a positive toxicology screen for opiates or cocaine
8. Prior history of diabetes mellitus
9. Prior history of chronic obstructive pulmonary disease (COPD) or asthma that is not clinically controlled (have not required systemic corticosteroids in the past month)
10. Prior history of HIV, not controlled or on medication
11. Peripheral white blood cell count of less than 3000
12. Acute worsening (<7 days) in respiratory symptoms (such as change in cough frequency or sputum production, fever, dyspnea, abnormal chest radiograph), or room air pulse oximetry of < 92% at rest or spirometry of < 50% predicted for FEV1 and FVC
13. Use of systemic antibiotics in the past month (4 weeks)
14. Failure of a subject or the subject's substance abuse counselor to provide assent
15. Nutritional risk index of less than 95
16. Age < 21 or > 55
17. Pregnancy
18. Decisionally challenged
19. Prisoners.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults aged 18 to 55 who have been exposed to chronic cannabis smoking (without a history of tobacco smoking) and health, non-smoking controls.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-11-11 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in alveolar macrophage phagocytosis related to the use of cannabis | Baseline and at 18 hours
  Alveolar macrophage phagocytosis, secretion of pro-inflammatory cytokines, and cellular apoptosis, both at baseline, and after stimulation with pathogen-associated molecular patterns.
Evaluation of intrapulmonary oxidative stress indices in bronchalveolar lavage (BAL) | Baseline
  Intrapulmonary oxidative stress indices will be measured in both isolated alveolar macrophages (AM) and acellular epithelial lining fluid derived from bronchoalveolar lavage (BAL).
Assessment of Lung Function | Baseline
  Spirometry/Pulmonary function testing

CONTACTS AND LOCATIONS:
Overall Officials: Ellen L Burnham, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Denver, Aurora, Colorado, United States